CLINICAL TRIAL: NCT01682291
Title: Pre-hYpertension tReament With A coMbinatIon of Dietary Supplements and Life-style Modifications
Brief Title: Prehypertension and Dietary Supplements - The PYRAMIDS Study
Acronym: PYRAMIDS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Assistant Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 450-B/2012/D
Record Dates: First submitted 2012-09-05; First posted 2012-09-10 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Prehypertension
Keywords: Prehypertension; Life-style modifications; Dietary supplementation
MeSH Terms: conditions — Prehypertension | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Life-style modifications (Active Comparator): Lifestyle modifications will include:
  Weight loss of as little as 10 lbs (4.5 kg) Adoption of the Dietary Approaches to Stop Hypertension (DASH) eating plan Dietary sodium should be reduced to no more than 2.4 g of sodium per day Regular aerobic physical activity (at least 30 minutes per day)
  Interventions: Behavioral: Life-style modifications
- Dietary supplements (Active Comparator): Life-style modifications along with a novel combination of dietary supplements that includes: Allium sativum (Dosage: 1,000 mg/day), Crataegus monogyna (Dosage: 500 mg/day), Orthosiphon (Dosage: 300 mg/day), Hibiscus sabdariffa (Dosage: 250 mg/day)
  Interventions: Dietary Supplement: Dietary supplements

INTERVENTIONS:
Behavioral: Life-style modifications — Weight loss of as little as 10 lbs (4.5 kg) Adoption of the Dietary Approaches to Stop Hypertension (DASH) eating plan Dietary sodium should be reduced to no more than 2.4 g of sodium per day Regular aerobic physical activity (at least 30 minutes per day)
  Other Names: Adoption of healthy lifestyles
  Arms: Life-style modifications
Dietary Supplement: Dietary supplements — combined pill (1 capsule/day containing Allium sativum (Dosage: 1,000 mg/day), Crataegus monogyna (Dosage: 500 mg/day), Orthosiphon (Dosage: 300 mg/day), Hibiscus sabdariffa (Dosage: 250 mg/day)
  Other Names: Life-style modifications and dietary supplements
  Arms: Dietary supplements

SUMMARY:
The primary objective of this study is to compare the efficacy and tolerability of a life-style modifications protocol versus a protocol including life-style modifications along with a novel combination of dietary supplement in the management of subjects diagnosed as having pre-hypertension.

The novel formulation includes: Allium sativum (Dosage: 1,000 mg/day), Crataegus monogyna (Dosage: 500 mg/day), Orthosiphon (Dosage: 300 mg/day), Hibiscus sabdariffa (Dosage: 250 mg/day)

DETAILED DESCRIPTION:
Prehypertension. Prehypertension is an American classification for those subjects with a normal-elevated blood pressure (BP) that does not reach the level considered to be hypertension.

Because of the new data on lifetime risk of hypertension and the impressive increase in the risk of cardiovascular complications associated with levels of BP previously considered to be normal, the JNC 7 report has introduced a new classification that includes the term "prehypertension" for those with BPs ranging from 120-139 mmHg systolic and/or 80-89 mmHg diastolic.

This new designation is intended to identify those individuals in whom early intervention by adoption of healthy lifestyles could reduce BP, decrease the rate of progression of BP to hypertensive levels with age, or prevent hypertension entirely.

Data from the 1999 and 2000 National Health and Nutrition Examination Survey (NHANES III) estimated that the prevalence of prehypertension among adults in the United States was approximately 31%. The prevalence is higher among men than women (39 and 23 percent, respectively).] People with prehypertension are at a higher risk for developing hypertension and target organ damages (i.e. left ventricular hypertrophy), as compared to people with normal blood pressure. Furthermore, similar to hypertension, prehypertension can increase the risk for heart attacks, strokes, congestive heart failure, and renal failure. Researchers have found that a prehypertensive person is 3 times more likely to have a heart attack and 1.7 times more likely to have heart disease than a person with normal blood pressure.

Management of Prehypertension.

* Prehypertension is not a disease category. Rather, it identifies individuals at high risk of developing hypertension, so that both patients and clinicians are alerted to this risk and encouraged to intervene and prevent or delay the disease from developing.
* Individuals who are prehypertensive are not candidates for drug therapy based on their level of BP and should be firmly and unambiguously advised to practice lifestyle modification in order to reduce their risk of developing hypertension.
* Moreover, individuals with prehypertension, who also have diabetes or kidney disease, should be considered candidates for appropriate drug therapy if a trial of lifestyle modification fails to reduce their BP to 130/80 mmHg or less.

Lifestyle Modifications. The goal for individuals with prehypertension and no compelling indications is to lower BP to normal levels with lifestyle changes, and prevent the progressive rise in BP using the recommended lifestyle modifications.

Also, adoption of healthy lifestyles is an indispensable part of the management of those with hypertension.

Lifestyle modifications include:

* Weight loss of as little as 10 lbs (4.5 kg) reduces BP and/or prevents hypertension
* Adoption of the Dietary Approaches to Stop Hypertension (DASH) eating plan94 which is a diet rich in fruits, vegetables, and low fat dairy products
* Dietary sodium should be reduced to no more than 100 mmol per day (2.4 g of sodium).
* Regular aerobic physical activity such as brisk walking at least 30 minutes per day
* Alcohol intake should be limited

Dietary Approaches to Stop Hypertension. The first-line approach to hypertension refractory to lifestyle modification remains pharmacologic therapy in combination with the low-salt DASH diet. However, a wide variety of alternative therapies are available for using to improve BP control. Dietary supplements and modification, as well as herbal supplements, may be useful under the right circumstances. Unfortunately, the efficacy of adding dietary, herbal, or alternative therapies is not well established. While combinations of antihypertensive drugs from different classes is a recommended approach that results in an additive benefit, it is not clear whether combinations of herbal or dietary supplements will also be additive.

Many of the studies evaluating the supplements referenced here are small and data are often derived from pooled analysis. In particular, studies to date evaluating garlic as well as many of the alternative approaches have significant limitations in study design. Should they prove efficacious and safe their use as a first-line therapy may come into play Thus, it remains unknown, however, whether the use of dietary supplements in association with life style interventions has any additive effect in subjects with Pre-hypertension.

Purpose The primary objective of this study is to compare the efficacy and tolerability of a life-style modifications protocol versus a protocol including life-style modifications along with a novel combination of dietary supplement in the management of subjects diagnosed as having pre-hypertension.

The novel formulation includes: Allium sativum (Dosage: 1,000 mg/day), Crataegus monogyna (Dosage: 500 mg/day), Orthosiphon (Dosage: 300 mg/day), Hibiscus sabdariffa (Dosage: 250 mg/day)

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy subjects with "prehypertension", that is blood pressures ranging from 120-139 mmHg systolic and/or 80-89 mmHg diastolic-

Exclusion Criteria:

* Women of child bearing potential patients must demonstrate a negative pregnancy test performed within 24 hours before CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Changes in blood pressure levels as compared with baseline at 1 year | 1 year
  Changes in systolic and diastolic blood pressure levels as compared with baseline at 1 year

SECONDARY OUTCOMES:
Reasons for treatment discontinuation | 1 year
  Reasons for treatment discontinuation during the 1-year study period

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Pelliccia, MD, Principal Investigator — Sapienza University
Locations (1):
- Sapienza University, Rome, Italy

REFERENCES:
- [Derived] Pelliccia F, Pasceri V, Marazzi G, Arrivi A, Cacciotti L, Pannarale G, Speciale G, Greco C, Gaudio C. Randomised, double-blind, placebo-controlled, assessment of the efficacy and safety of dietary supplements in prehypertension. J Hum Hypertens. 2017 Oct;31(10):647-653. doi: 10.1038/jhh.2017.35. Epub 2017 Apr 27. PMID 28447625